CLINICAL TRIAL: NCT02069119
Title: A Multicenter, Parallel-group-comparison, Double-blind, Placebo-controlled, Randomized Trial to Determine the Safety, Pharmacokinetics, and Efficacy of OPC-108459 Administered as a Single Intravenous Dose to Patients With Paroxysmal or Persistent Atrial Fibrillation
Brief Title: A Trial to Determine the Safety, Pharmacokinetics, and Efficacy of OPC-108459 Administered as a Single Intravenous Dose to Patients With Paroxysmal or Persistent Atrial Fibrillation (AF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 269-13-001
Record Dates: First submitted 2014-02-20; First posted 2014-02-21 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- OPC-108459 (Experimental): OPC-108459 solution will be intravenously administered by 30-minute infusion in the forearm.
  Interventions: Drug: OPC-108459
- Placebo (Placebo Comparator): placebo solution will be intravenously administered by 30-minute infusion in the forearm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPC-108459
  Arms: OPC-108459
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate the safety, pharmacokinetics, and efficacy following 30-minute continuous intravenous administration of OPC-108459 at 0.4, 0.8, 1.6, or 2.4 mg/kg or placebo to patients with paroxysmal or persistent atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

* Japanese
* Male or female age 20 to 85 years, inclusive (at the time of informed consent)
* Patients diagnosed with recent or new onset of paroxysmal AF (3 hours to 7 days since the onset) or persistent AF (8 to 30 days since the onset) at time of randomization (prior to Investigational Medicinal Product [IMP] administration). Review of the patient's medical records and the judgment of the investigator or sub-investigator must be documented in the source documents to establish the date and duration of the most recent onset of AF.
* Patients who are receiving treatment according to the "Guidelines for Pharmacotherapy of Atrial Fibrillation (JCS 2008)" at time of screening and predosing examinations or who have a low risk of thromboembolic potential specified as follows:

  * AF lasting less than 48 hours, OR
  * For AF lasting for 48 hours or longer:

    * Patients receiving warfarin therapy for whom at least 3 weeks have elapsed since achieving an international normalized ratio (INR) of 2.0 to 3.0 (1.6 to 2.6 for patients age 70 years or older) or in whom no thrombus in the atrial main body or appendage is observed by transesophageal echocardiography (TEE) within 24 hours before IMP administration
    * Patients in whom no thrombus in the atrial main body or appendage is observed by TEE within 24 hours before IMP administration if they have not undergone antithrombotic therapy or if they have undergone antithrombotic therapy (including a new oral antithrombotic drug) which does not meet the above criterion
* Patients with systolic blood pressure (sBP) of 90 mmHg or higher and lower than 160 mmHg and diastolic blood pressure (dBP) of lower than 100 mmHg at screening examinations
* Female patients who have been postmenopausal for at least 12 consecutive months, or male and female patients who agree, together with their partners, to practice birth control as specified until 3 months after the start of IMP administration or who are surgically sterile (ie, have undergone orchiectomy or hysterectomy, respectively)

Exclusion Criteria:

* QRS interval of > 120 msec
* Patients with heart failure of New York Heart Association (NYHA) Class II to IV or with left ventricular ejection fraction (LVEF) of < 40%
* Patients who currently have or have a history of a long QT syndrome, torsade de pointes, or an uncorrected QT interval of > 450 msec
* History of ventricular tachycardia, ventricular fibrillation, or resuscitated cardiac arrest
* History of AF and failed electrical or pharmacological cardioversion
* Current diagnosis of atrial flutter
* Patients with bradycardia (< 50 beats per minute [bpm]) or sick sinus syndrome, unless controlled by a pacemaker, except for physiologically transient sinus bradycardia observed at rest or during sleep
* Patients with Wolff-Parkinson-White syndrome
* Patients with any congenital severe heart disease
* Patients with severe aortic or mitral stenosis (aortic-valve area, < 1 cm2), severe mitral regurgitation, aortic regurgitation, congenital atrial septal defect, moderate or severe pulmonary hypertension, or any other disease leading to AF confirmed by echocardiography within one year prior to screening examinations
* Patients diagnosed with congenital valvular anomaly or severe valve disease (eg, aortic or mitral stenosis, severe right or left ventricular systolic dysfunction, or severe pulmonary hypertension) and confirmed current presence of the condition by TEE at screening examinations
* Patients diagnosed with stroke or transient ischemic attack within one year prior to screening examinations or with carotid artery stenosis of 50%
* History of myocardial infarction within 6 months prior to screening examinations
* Findings of acute coronary syndrome, angina, or myocardial ischemia diagnosed by ECG or drug-induced or exercise stress testing within 6 months prior to screening examinations

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kyushu Region, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- OPC-108459（Paroxysmal AF）; OPC-108459 (Persistent AF): Randomized: 20/24 subjects
- Placebo（Paroxysmal AF）; Placebo (Persistent AF）: Randomized: 4/24 subjects
Period: Overall Study
Arm/Group | OPC-108459（Paroxysmal AF） | Placebo（Paroxysmal AF） | OPC-108459 (Persistent AF) | Placebo (Persistent AF）
Started | 20 | 4 | 20 | 4
Completed | 20 | 4 | 20 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-108459（Paroxysmal） | Placebo（Paroxysmal） | OPC-108459（Persistent） | Placebo（Persistent） | Total
Number analyzed (Participants) | 20 | 4 | 20 | 4 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 9 | 3 | 16
  >=65 years | 17 | 3 | 11 | 1 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (7.7) | 67.5 (3.8) | 65.4 (8.8) | 60.0 (13.3) | 67.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 7 | 0 | 16
  Male | 13 | 2 | 13 | 4 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 20 | 4 | 20 | 4 | 48

OUTCOME MEASURES:

1. Primary Outcome: Subjects Achieving Normal Sinus Rhythm (NSR) in Patients With Paroxysmal AF
Description: 24 subjects with paroxysmal AF, 6 subjects per cohort (5 for OPC-108459 and one for placebo), 4 dose steps; Step 1: 0.4 mg/kg, Step 2: 0.8 mg/kg, Step 3: 1.6 mg/kg, Step 4: 2.6 mg/kg
  The number of subjects achieving NSR within 90 minutes after the start of IMP administration and sustaining NSR for at least one minute.
Time Frame: 90 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | OPC-108459 Step 1 (0.4 mg/kg) | OPC-108459 Step 2 （0.8 mg/kg） | OPC-108459 Step 3 （1.6mg/kg） | OPC-108459 Step 4 （2.6 mg/kg） | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 4
Participants | 0 | 2 | 0 | 0 | 0

2. Primary Outcome: Subjects Achieving NSR in Patients With Persistent AF
Description: 24 subjects with persistent AF, 6 subjects per cohort (5 for OPC-108459 and one for placebo), 4 dose steps; Step 1: 0.4 mg/kg, Step 2: 0.8 mg/kg, Step 3: 1.6 mg/kg, Step 4: 2.6 mg/kg
  The number of subjects achieving NSR within 90 minutes after the start of IMP administration and sustaining NSR for at least one minute.
  No subjects achieved NSR within 90 minutes after the start of IMP administration in the persistent AF cohort.
Time Frame: 90 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | OPC-108459 Step 1 (0.4 mg/kg) | OPC-108459 Step 2 （0.8 mg/kg） | OPC-108459 Step 3 （1.6mg/kg） | OPC-108459 Step 4 （2.6 mg/kg） | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 4
Participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Cmax of Plasma OPC-108459 in Patients With Paroxysmal AF
Description: Of 20 subjects for whom plasma OPC-108459 concentrations were measured, 19 subjects were included in the PK analysis, and one subject was excluded.
Time Frame: 0, 30, 50 minute and 2, 4, 8, 24 hour
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OPC-108459 Step 1 （0.4 mg/kg） | OPC-108459 Step 2 （0.8 mg/kg） | OPC-108459 Step 3 （1.6mg/kg） | OPC-108459 Step 4 （2.6 mg/kg）
Number analyzed (Participants) | 5 | 5 | 5 | 4
ng/mL | 786.2 (228.1) | 1942.0 (2428.0) | 3629.0 (499.1) | 5316.0 (1230.0)

4. Primary Outcome: Cmax of Plasma OPC-108459 in Patients With Persistent AF
Description: Of 20 subjects for whom plasma OPC-108459 concentrations were measured, all subjects were included in the PK analysis.
Time Frame: 0, 30, 50 minute and 2, 4, 8, 24 hour
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OPC-108459 Step 1 （0.4 mg/kg） | OPC-108459 Step 2 （0.8 mg/kg） | OPC-108459 Step 3 （1.6mg/kg） | OPC-108459 Step 4 （2.6 mg/kg）
Number analyzed (Participants) | 5 | 5 | 5 | 5
ng/mL | 1037.0 (154.5) | 1593.0 (382.1) | 3676.0 (826.8) | 6412.0 (964.6)

ADVERSE EVENTS:
Time Frame: From the start date of IMP administration to date of the final examination (up to 30 days after IMP administration)
Groups:
- OPC-108459（Paroxysmal）; Placebo（Paroxysmal）: A total of 112 subjects were enrolled and screened, and 48 subjects were randomized to either the OPC-108459 group or placebo group. Of the 48 subjects, 24 subjects were randomized to paroxysmal AF cohort (20 for the OPC-108459, 4 for the placebo). All the randomized subjects received the Interventional medicinal product (IMP) administration and were included in the FAS. Of the 24 subjects, 18 subjects were included in the PK analysis set.
- OPC-108459（Persistent）; Placebo（Persistent）: Of the 48 subjects, 24 subjects were randomized to persistent AF cohort (20 for the OPC-108459, 4 for the placebo). All the randomized subjects in Persistent AF cohort received the IMP administration and were included in the FAS and PK analysis set.
Arm/Group | OPC-108459（Paroxysmal） | OPC-108459（Persistent） | Placebo（Paroxysmal） | Placebo（Persistent）
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 9/20 | 12/20 | 2/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-108459（Paroxysmal） (N=20) | OPC-108459（Persistent） (N=20) | Placebo（Paroxysmal） (N=4) | Placebo（Persistent） (N=4)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-108459（Paroxysmal） (N=20) | OPC-108459（Persistent） (N=20) | Placebo（Paroxysmal） (N=4) | Placebo（Persistent） (N=4)
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Mydriasis (Eye disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 2 | 0 | 1 | 0
Atrial tachycardi (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Vascular pain (Vascular disorders) | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Chest discomfort (General disorders) | 1 | 1 | 1 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Blood pressure decreased (Investigations) | 3 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0
Glucose urine present (Investigations) | 1 | 2 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0
Heart rate increased1 (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram RR interval prolonged (Investigations) | 0 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0
Respiratory rate increased (Investigations) | 1 | 0 | 0 | 0
Heat illness (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No